CLINICAL TRIAL: NCT05794204
Title: A Phase 2a Study Evaluating the Safety and Efficacy of RMP-A03 Ocular Suspension in Patients With Pterygium
Brief Title: RMP-A03 Ocular Suspension in Patients With Pterygium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Raymon Pharmaceuticals Company, Ltd. (Industry)
Collaborators: WuXi Clinical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RMP-A03-001
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1:1 fashion
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor/CRO clinical operations team will also be masked. Sponsor/CRO biostats team and drug supply manager will be unmasked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Patients randomized to dose 1 study drug (Experimental): Approximately 25 patients randomized to dose 1 of RMP-A03
  Interventions: Drug: RMP-A03 - Dose 1
- Patients randomized to dose 2 of study drug (Experimental): Approximately 25 patients randomized to dose 2 of RMP-A03
  Interventions: Drug: RMP-A03 - Dose 2
- Patients randomized to placebo (Placebo Comparator): Approximately 25 patients randomized to placebo.
  Interventions: Drug: RMP-A03 Placebo

INTERVENTIONS:
Drug: RMP-A03 - Dose 1 — Patients will randomized to low dose of RMP-A03
  Arms: Patients randomized to dose 1 study drug
Drug: RMP-A03 - Dose 2 — Patients will be randomized to high dose of RMP-A03
  Arms: Patients randomized to dose 2 of study drug
Drug: RMP-A03 Placebo — Patients will be randomized to RMP-A03 Placebo
  Arms: Patients randomized to placebo

SUMMARY:
The goal of this clinical trial is to test the safety and efficacy of an ocular medication on the treatment of pterygium.

DETAILED DESCRIPTION:
Following informed consent, patients with pterygium who meet all eligibility criteria will be randomized to an 84-day double-blinded study to measure the safety and efficacy of the study drug as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years old
* Diagnosis of pterygium with specified characteristics
* BCVA of 20/200 or better
* Willingness to attend all study visits and comply with the study procedures

Exclusion Criteria:

* Presence of ocular disease
* Double pterygium
* History of ocular surgery
* Presence of ocular trauma
* Use of any ocular medication
* Use of contact lens
* Allergy to any of the components of study drug
* Cannot properly administer study drug
* Clinically significant systemic disease that may place the subject at risk or confound study results
* Participation in an investigational study within 30 days prior to screening
* Female participants who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control (WOCBP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pterygium hyperemia grading at Day 28 | 28 days
  Pterygium hyperemia grading will be assessed by the principal investigator based on predefined vascularity scale.

SECONDARY OUTCOMES:
Change from baseline in pterygium characteristics at Day 28 | 28 days
  Pterygium size will be measured by the principal investigator based on predefined scale

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Global Research Management, Glendale, California
  - United Medical Research Institute, Inglewood, California
  - Eye Research Foundation Inc, Newport Beach, California
  - Oceane7 Medical & Research Center Inc., Miami, Florida
  - Toyos Clinic, Nashville, Tennessee
  - Keystone Research, Austin, Texas